CLINICAL TRIAL: NCT01185782
Title: Parallel-Group Comparative Study of SJ-0021 and Purified Pituitary Gonadotropin in Subjects With Amenorrhea I or Anovulatory Cycles - Phase III Single-Blind Study
Brief Title: SJ-0021 (Gonalef®) Versus Purified Pituitary Gonadotropin (Fertinorm-P®) for Ovulation Induction in Japanese Infertile Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Co., Ltd., Japan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMP26648; NCT00467480 (obsolete NCT alias)
Record Dates: First submitted 2010-08-11; First posted 2010-08-20 (Estimated); Results first posted 2012-02-24 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Infertility; Ovulation Induction
Keywords: Infertility; Ovulation induction; Gonalef® (Follitropin alfa); Purified pituitary gonadotropin (Fertinorm-P®); gonadotropin; Reproductive technologies, assisted; Polycystic ovary syndrome
MeSH Terms: conditions — Infertility; Helping Behavior; Polycystic Ovary Syndrome | interventions — follitropin alfa; Urofollitropin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SJ-0021 group (Experimental)
  Interventions: Drug: Gonalef® (Follitropin alfa)
- Purified pituitary gonadotropin group (Active Comparator)
  Interventions: Drug: Purified pituitary gonadotropin (Fertinorm-P®)

INTERVENTIONS:
Drug: Gonalef® (Follitropin alfa) — Subcutaneous administration of follitropin alfa at a dose of 75 IU/day was started on dosing Day 1 and the same daily dose was maintained for the first 7 days of the treatment period. Dose increment by 37.5 IU was permitted on dosing Day 8, Day 15 and Day 22 if the dosage increase criterion was met.
  Other Names: Gonalef®; follitropin alfa; recombinant human follicle-stimulating hormone; r-hFSH; SJ-0021
  Arms: SJ-0021 group
Drug: Purified pituitary gonadotropin (Fertinorm-P®) — Subcutaneous administration of purified pituitary gonadotropin at a dose of 75 IU/day was started on dosing Day 1 and the same daily dose was maintained for the first 7 days of the treatment period. Dose increment by 37.5 IU was permitted on dosing Day 8, Day 15 and Day 22 if the dosage increase criterion was met.
  Other Names: Fertinorm-P®; purified urinary human follicle-stimulatin hormone; urofollitropin; u-hFSH
  Arms: Purified pituitary gonadotropin group

SUMMARY:
Efficacy and safety studies in the past have suggested that a starting dose of 75 International Unit (IU) of SJ-0021, and an increase in the dose by 37.5 IU every 7 days, are safe for treatment of subjects with ovulatory disorders who are infertile due to hypothalamic or pituitary dysfunction and have amenorrhea I or anovulatory cycles (including oligomenorrhea and polymenorrhea).

This was a phase III, multicentre, single-blind, parallel-group comparative study conducted to provide confirmatory evidence of non-inferiority of SJ-0021 versus purified gonadotropin, a comparator drug, for induction of follicle development and ovulation in infertile Japanese women and to provide further information on the safety and tolerability of SJ-0021.

DETAILED DESCRIPTION:
Follicle stimulating hormone (FSH) is a heterodimeric glycoprotein wherein an alfa subunit and a beta subunit are noncovalently bonded. Follicle stimulating hormone is one of the key hormones regulating reproductive functions in both female and male mammals, including humans. In females, it stimulates the development of ovarian follicles, which carry oocytes, while in males it promotes spermatogenesis. Synthesis and secretion of FSH are stimulated by gonadotropin releasing hormone (GnRH), a hypothalamic peptide. Complete or partial deficiencies in FSH secretion are common causes of infertility in men and women. In women, this state is characterized by absence of ovulation or abnormal ovulation. In men, it leads to absence of or abnormally low production of spermatozoa. Administration of FSH, either alone or in combination with luteinizing hormone (LH), has been used successfully to treat these infertility problems. Until recently, only human menopausal gonadotropin (hMG), a mixture of human LH and FSH extracted from the urine of post-menopausal women, and purified FSH (u-hFSH), which could be used to reduce the LH content, had been available for treatment of infertility. In Japan, hMG and u-hFSH are still used to induce ovulation.

Purified pituitary gonadotropin, which was used as the comparator drug in this clinical trial, is a urinary gonadotropin preparation. However, it is not classified as hMG, but rather as a purified pituitary gonadotropin (u-hFSH), and is the preparation most commonly used in Japan. Since the LH content of u-hFSH is very low, it can be administered relatively safely, if adequate care is taken, to patients with polycystic ovary syndrome (PCOS). SJ-0021 is a recombinant human FSH (r-hFSH) that is produced using Chinese hamster ovary (CHO) cells as the host cells. The generic name for SJ-0021 is follitropin alfa for injection, and it is marketed overseas as GONAL-f®. It was approved in Japan in January 2006 as being effective in inducing spermatogenesis in cases of male hypogonadotropic hypogonadism (MHH).

OBJECTIVES

* To examine the efficacy of SJ-0021 versus purified pituitary gonadotropin for ovulation induction and follicle development in subjects with amenorrhea I or anovulatory cycles, and to verify the non-inferiority of SJ-0021 versus the comparator drug
* To assess the safety of SJ-0021

This clinical trial comprised of a pretrial observation period, a treatment period [IMP administration period], and a post-treatment assessment period. The clinical trial was scheduled in such a way that spontaneous menstruation or withdrawal bleeding induced by progesterone administration occurred within 28 days after the completion of baseline tests conducted during the pretrial observation period. A visit to the trial site was then scheduled for any day between Day 2-5 of the spontaneous menstruation or withdrawal bleeding, during which actual registration of the subject for randomization and pre-administration tests were performed. After completion of pre-administration tests, 75 IU of either SJ-0021 or purified pituitary gonadotropin that was allocated to the subject was subcutaneously administered on the same day (dosing Day 1 of treatment period), and the same daily dose was maintained for the first 7 days of the treatment period. On dosing Day 8, the mean diameter of the dominant follicle was measured; if it was < 11 mm, the daily IMP dose was increased by 37.5 IU and this new daily dose was administered for the next 7 days. If the mean diameter of the dominant follicle was ≥ 11 mm but < 18 mm, the same (previous) IMP dose was administered for the next 7 days. If the mean diameter of the dominant follicle had already reached 18 mm or above, administration of the IMP was terminated, and the subject moved on to the post treatment assessment period. Similarly, if the mean diameter of the dominant follicle was < 11 mm on dosing Day 15 or Day 22, the dose was increased; if it was ≥ 11 mm but < 18 mm, administration was continued at the same previous dose, and if it was ≥ 18 mm IMP administration was terminated. The maximum dose of IMP that can be administered was 187.5 IU/day and the maximum dosing period for the IMP was 28 days. In addition to Day 8, Day 15 and Day 22, ultrasound examination can be conducted once or twice a week during the treatment period, based on the status of growth of the dominant follicle (and on every visit once the dominant follicle has achieved a maximum diameter of 16 mm).

Examinations for the first day of the post-treatment assessment period were conducted, as appropriate, on the day when the mean diameter of the dominant follicle reached ≥ 18 mm or on the day after dosing Day 28 of the IMP. The hCG cancellation criterion (i.e. four or more ovarian follicles with a mean diameter ≥ 16 mm) was also verified at the same time. If the hCG cancellation criterion was not met, a single dose of 5000 IU of hCG was administered intramuscularly, within 24 hours of the last ultrasound examination. Mid-luteal phase tests were conducted on Day 6 ± 1 and Day 9 ± 1 of the post-treatment assessment period, and a final examination was performed on Day 28-31 of the post-treatment assessment period. If the pregnancy test (urine) conducted at this final examination was positive, a further pregnancy test (ultrasound examination) was performed on Day 35-42 of the post-treatment assessment period.

On the other hand, if the mean diameter of the dominant follicle remained < 16 mm on the day after dosing Day 28 of the IMP, or the hCG cancellation criterion was met, hCG administration was withheld, and the examinations for the first day of the post-treatment assessment period as well as the final examination on Day 28-31 of the post-treatment assessment period were performed accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20 to 39 years (inclusive) who hope to bear children
* Subjects who failed to achieve ovulation or pregnancy despite 2 cycles or more of anti-estrogen therapies (clomiphene citrate, cyclofenil, etc.)
* Subjects who exhibited withdrawal bleeding in a progesterone test (Includes spontaneous menstruation in subjects with anovulatory cycles.)
* Subjects having a body mass index between 17.0 and 28.0 at the time of baseline tests
* Subjects who voluntarily consented in writing to participate in the clinical trial

Exclusion Criteria:

* Subjects with ovarian tumors
* Subjects with ovarian enlargement not due to PCOS
* Subjects with genitourinary hemorrhage of unknown cause
* Subjects who were or may be pregnant, or who were lactating
* Subjects with history of allergic reaction or hypersensitivity to gonadotropin
* Subjects with dysfunction of heart, lungs, kidneys, or cardiovascular systems of Grade 2 or higher (in compliance with the Pharmaceutical and Medical Safety Bureau Notification Yakuan No. 80 [issued 29 June 1992])
* Subjects with serum progesterone (P4) level ≥ 5 ng/mL in baseline tests
* Subjects with malignant tumors
* Subjects with uterine amenorrhea
* Subjects with elevated levels of serum gonadotropin due to premature ovarian failure (FSH ≥ 20 mIU/mL)
* Subjects who were infertile due to known adrenal or thyroid dysfunction
* Subjects who were diagnosed as having hyperprolactinemia
* Subjects who had been documented or suspected of having intracranial lesions (e.g., pituitary tumors)
* Infertile subjects involving gynecological factors other than amenorrhea I or anovulatory cycles, and for whom ovulation induction therapy was found to be contraindicated
* Subjects who had participated in another clinical study within 6 months prior to start of the IMP administration
* Subjects who had been administered SJ-0021 in the past
* Subjects whose participation in this clinical trial was otherwise deemed inappropriate by the investigator or sub-investigator

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2007-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimitoshi Takemura, Study Director — Merck Serono Co., Ltd., Japan
Locations (1):
- The University of Tokyo Hospital, Tokyo, Japan

REFERENCES:
- [Result] Taketani Y, Kelly E, Yoshimura Y, Hoshiai H, Irahara M, Mizunuma H, Saito H, Andoh K, Yanaihara T. Recombinant follicle-stimulating hormone (follitropin alfa) versus purified urinary follicle-stimulating hormone in a low-dose step-up regimen to induce ovulation in Japanese women with anti-estrogen-ineffective oligo- or anovulatory infertility: results of a single-blind Phase III study. Reprod Med Biol. 2010 Feb 23;9(2):99-106. doi: 10.1007/s12522-010-0046-5. eCollection 2010 Jun. PMID 29699333

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in 21 study centers in Japan from 15 February 2007 to 25 December 2007.
Pre-assignment Details: 300 participants were enrolled in the study; 39 participants discontinued prior to Investigational Medicinal Product (IMP) administration (35 participants for no longer meeting the eligibility criteria 4 due to Adverse Events [AEs] or other reasons). Demographic data was not available for the 4 participants who were randomized but not treated.
Groups:
- SJ-0021: SJ-0021 (recombinant follitropin alfa) was administered subcutaneously (s.c.) at a starting dose of 75 International Unit (IU)/day which was to be followed by incremental doses of 37.5 IU on Days 8, 15 and 22 if the mean dominant follicle diameter was less than 11 mm. The maximum duration of treatment was 28 days.
- u-hFSH: Urinary human follicle stimulating hormone (u-hFSH), a purified pituitary gonadotropin, was administered s.c. at a starting dose of 75 IU/day which was to be followed by incremental doses of 37.5 IU on Days 8, 15 and 22 if the mean dominant follicle diameter was less than 11 mm. The maximum duration of treatment was 28 days.
Period: Overall Study
Arm/Group | SJ-0021 | u-hFSH
Started | 129 | 136
Treated | 129 | 132
Completed | 123 | 125
Not Completed | 6 | 11
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Poor Response to Treatment | 3 | 1
Not completed — Other | 2 | 5
Not completed — Randomized but not treated | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SJ-0021 | u-hFSH | Total
Number analyzed (Participants) | 129 | 132 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (3.8) | 31.6 (3.8) | 31.6 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 132 | 261
  Male | 0 | 0 | 0
Previous episodes of Ovarian hyperstimulation syndrome (OHSS) [Number; unit: participants] — OHSS is a syndrome which can manifest with enlarged ovaries, advanced ascites with increased vascular permeability, pleural fluid accumulation, hemoconcentration, and increased blood clotting. Episodes of OHSS are presented as values from 0 to 4 where 0 = no episodes to 4 = four episodes.
  participants
    0 | 116 | 119 | 235
    1 | 9 | 10 | 19
    2 | 2 | 3 | 5
    3 | 1 | 0 | 1
    4 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Ovulation
Description: Participants were considered to have ovulated if serum progesterone (P4) level was greater than or equal to 5 nanogram (ng)/mL on Day 6±1 or 9±1 during the post-treatment assessment period, or if the participant became clinically pregnant.
Time Frame: On Day 6±1 or 9±1 days during post-treatment assessment period (Day 35-42 of post-treatment period for clinical pregnancy)]
Population: Full analysis set (FAS) included all participants who received at least 1 dose of IMP and had no major violation of Good Clinical Practice (GCP) such as non-compliance with the agreement, serious protocol violations, etc.
Measure: Number; unit: percentage of participants
Arm/Group | SJ-0021 | u-hFSH
Number analyzed (Participants) | 129 | 132
percentage of participants | 79.1 | 82.6
Statistical Analysis 1: Comparison: SJ-0021 vs u-hFSH; Test type: Non-Inferiority or Equivalence — The primary endpoint was to determine whether or not SJ-0021 is inferior to u-hFSH in inducing ovulation. The criterion for non-inferiority was that the lower limit of the two-sided 95% CI (= one-sided 97.5% CI) had to be greater than -15% for SJ-0021 to be considered not inferior to u-hFSH."); Chi-squared; Delta = -3.51, 95% CI 2-sided [-13.05 to 6.04]

2. Secondary Outcome: Number of Participants With the Dominant Follicle Achieving 18 mm in Mean Diameter
Time Frame: Start of treatment period until Day 1 of post-treatment assessment period
Population: FAS included all participants who received at least 1 dose of IMP and had no major violation of GCP such as non-compliance with the agreement, serious protocol violations, etc.
Measure: Number; unit: participants
Arm/Group | SJ-0021 | u-hFSH
Number analyzed (Participants) | 129 | 132
participants | 117 | 125
Statistical Analysis 1: Comparison: SJ-0021 vs u-hFSH; Test type: Superiority or Other; p = 0.214, Chi-squared

3. Secondary Outcome: Time for Dominant Follicle to Achieve 18 mm in Mean Diameter
Description: Dosing time length was calculated as number of days from the first administration of the IMP until the mean diameter of the dominant follicle was confirmed to have reached 18 mm.
Time Frame: Start of treatment period until Day 1 of post-treatment assessment period
Population: FAS included all participants who received at least 1 dose of IMP and had no major violation of GCP such as non-compliance with the agreement, serious protocol violations, etc. Only participants in whom the dominant follicle reached 18 mm in mean diameter were considered for the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | SJ-0021 | u-hFSH
Number analyzed (Participants) | 117 | 125
days | 13.1 (5.1) | 12.1 (4.2)
Statistical Analysis 1: Comparison: SJ-0021 vs u-hFSH; Test type: Superiority or Other; p = 0.087, t-test, 2 sided

4. Secondary Outcome: Total Dose of the Investigational Medicinal Product (IMP) Administered to Participants With Dominant Follicle Achieving 18 mm in Mean Diameter
Description: Total dose of IMP administered was defined as the cumulative dose administered from the start of treatment with IMP until the mean diameter of the dominant follicle reached 18 mm.
Time Frame: Start of treatment period until Day 1 of post-treatment assessment period
Population: FAS included all participants who received at least 1 dose of IMP and had no major violation of GCP such as non-compliance with the agreement, serious protocol violations, etc. Only participants in whom the dominant follicle reached 18 mm in mean diameter were considered for the analysis of this parameter.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | SJ-0021 | u-hFSH
Number analyzed (Participants) | 117 | 125
IU | 959.29 (533.32) | 845.70 (432.88)
Statistical Analysis 1: Comparison: SJ-0021 vs u-hFSH; Test type: Superiority or Other; p = 0.069, t-test, 2 sided

5. Secondary Outcome: Human Chorionic Gonadotropin (hCG) Cancellation Rate
Description: hCG cancellation criterion was defined as the presence of 4 or more ovarian follicles with a mean diameter greater than or equal to 16 mm. If the hCG cancellation criterion was met, the administration of hCG was withheld. Otherwise, a single intramuscular dose of hCG 5000 IU (Japanese Pharmacopoeia- JP) was administered within 24 hours of the last ultrasound examination.
Time Frame: Day 1 of post-treatment assessment period
Population: as for outcome 2
Measure: Number; unit: percent hCG cancellation
Arm/Group | SJ-0021 | u-hFSH
Number analyzed (Participants) | 129 | 132
percent hCG cancellation | 7.0 | 7.6
Statistical Analysis 1: Comparison: SJ-0021 vs u-hFSH; Test type: Superiority or Other; p = 0.852, Chi-squared

6. Secondary Outcome: Single Follicle Maturation Rate
Description: Single follicle maturation was defined as the presence of the dominant follicle with a mean diameter of 18 mm or greater without concurrent presence of other follicles of 14 mm or larger in diameter.
Time Frame: Start of treatment period until Day 1 of post-treatment assessment period
Population: as for outcome 2
Measure: Number; unit: percent single follicle maturation
Arm/Group | SJ-0021 | u-hFSH
Number analyzed (Participants) | 129 | 132
percent single follicle maturation | 33.3 | 43.2
Statistical Analysis 1: Comparison: SJ-0021 vs u-hFSH; Test type: Superiority or Other; p = 0.102, Chi-squared

7. Secondary Outcome: Biochemical Pregnancy Rate
Description: Biochemical pregnancy was defined as a positive pregnancy test (urinary beta-hCG test) on Day 28-31 of the post-treatment assessment period
Time Frame: Day 28-31 of post-treatment assessment period
Population: as for outcome 2
Measure: Number; unit: percent biochemical pregnancy
Arm/Group | SJ-0021 | u-hFSH
Number analyzed (Participants) | 129 | 132
percent biochemical pregnancy | 17.8 | 15.2
Statistical Analysis 1: Comparison: SJ-0021 vs u-hFSH; Test type: Superiority or Other; p = 0.560, Chi-squared

8. Secondary Outcome: Clinical Pregnancy Rate
Description: Clinical pregnancy was defined as existence of at least one ultrasonography confirmed gestational sac in the uterus, with or without heartbeat.
Time Frame: Day 35-42 of post-treatment assessment period
Population: as for outcome 2
Measure: Number; unit: percent clinical pregnancy
Arm/Group | SJ-0021 | u-hFSH
Number analyzed (Participants) | 129 | 132
percent clinical pregnancy | 17.1 | 14.4
Statistical Analysis 1: Comparison: SJ-0021 vs u-hFSH; Test type: Superiority or Other; p = 0.555, Chi-squared

9. Secondary Outcome: Ovulation Rate, Where Ovulation is Defined as a Serum P4 Level Greater Than or Equal to 10 ng/mL or Clinical Pregnancy
Description: For this secondary endpoint, participants were considered to have ovulated if serum P4 level was more than or equal to 10 ng/mL on Day 6±1 or 9±1 during the post-treatment assessment period, or if the participant became clinically pregnant.
Time Frame: On Day 6±1 or 9±1 during post-treatment assessment period
Population: as for outcome 2
Measure: Number; unit: percent ovulation
Arm/Group | SJ-0021 | u-hFSH
Number analyzed (Participants) | 129 | 132
percent ovulation | 71.3 | 75.8
Statistical Analysis 1: Comparison: SJ-0021 vs u-hFSH; Test type: Superiority or Other; p = 0.416, Chi-squared

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and AEs Leading to Study Drug Discontinuation
Description: AEs: Any untoward medical occurrence in the form of signs, clinically significant abnormalities in laboratory findings, diseases, symptoms, or worsening of complications. TEAEs: AEs that occur during treatment with the IMP. SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was a medically important condition. Participants who discontinued from the study due to AE were also recorded.
Time Frame: Pretrial observation period to post-treatment assessment period (Days 35-42)
Population: Safety population included all participants who received at least 1 dose of IMP. This was actually identical to the FAS population.
Measure: Number; unit: participants
Arm/Group | SJ-0021 | u-hFSH
Number analyzed (Participants) | 129 | 132
participants
  TEAEs | 69 | 66
  SAEs | 1 | 1
  Discontinuation due to AEs | 0 | 1

11. Secondary Outcome: Number of Participants With OHSS
Description: OHSS is a syndrome which can manifest with enlarged ovaries, advanced ascites with increased vascular permeability, pleural fluid accumulation, hemoconcentration, and increased blood clotting.
Time Frame: Start of treatment period to post-treatment assessment period (Day 35-42)
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | SJ-0021 | u-hFSH
Number analyzed (Participants) | 129 | 132
participants | 10 | 5

ADVERSE EVENTS:
Time Frame: AEs were collected on an ongoing basis from day of written informed consent. All new AEs must be recorded until the final post-treatment examination, on Day 35-42 of the post-treatment assessment period.
Arm/Group | SJ-0021 | u-hFSH
Serious Adverse Events (participants affected / at risk) | 1/129 | 1/132
Other Adverse Events (participants affected / at risk) | 36/129 | 40/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SJ-0021 (N=129) | u-hFSH (N=132)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SJ-0021 (N=129) | u-hFSH (N=132)
Abdominal pain lower (Gastrointestinal disorders) | 6 (7) | 14 (17)
Abdominal distension (Gastrointestinal disorders) | 9 (10) | 7 (7)
Ascites (Gastrointestinal disorders) | 4 (4) | 7 (7)
Nasopharyngitis (Infections and infestations) | 10 (10) | 11 (11)
Headache (Nervous system disorders) | 6 (6) | 8 (9)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 9 (9) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other